CLINICAL TRIAL: NCT03379610
Title: A Prospective Study of Molecular Detection of Salvageable Early Recurrent Nasopharyngeal Carcinoma After Radiotherapy
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Dora Kwong, Clinical Professor, The University of Hong Kong
Other Study IDs: NP swabs
Record Dates: First submitted 2017-12-10; First posted 2017-12-20 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal brush NPC biopsy specimen Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nasopharngeal brush — 1. Baseline nasopharngeal brush before treatment
  2. Post-treatment reassessment of residual NPC
  Other Names: Nasopharngeal swabs

SUMMARY:
To evaluate the sensitivity and specificity of the combination of EBV and methylation marker genes in body fluids of both plasma and nasopharyngeal brush together for screening of early salvageable local residual and recurrent NPC that are missed by conventional clinical follow-up protocol.

DETAILED DESCRIPTION:
1. Background: Treatment failure can occur at distant sites which have no effective cure yet. Early local residual or recurrent NPC are salvageable with over 50% 5-year survival rate. It is however difficult for clinical detection of early residual or recurrent NPC after radiotherapy by nasoendoscopy in the heavily irradiated nasopharynx with severe nasopharyngitis and inflammatory swelling and crusting changes. Radiologic imaging and nasopharyngeal biopsy have their role, but they are invasive, expensive and cannot be repeated often as routine follow-up screening method. Unfortunately, 50% local recurrences are in advanced rT3-4 stage and 28% local recurrences are not salvageable. Therefore, detection of the early stage residual/recurrent NPC that are missed by our conventional clinical follow-up is important for successful salvage treatment. Non-invasive, inexpensive and repeatable sampling of blood and nasopharyngeal brush/swab for molecular detection of NPC is our research focus for future improvement of treatment result of local failure.

There are two potential molecular markers of detection of minimal residual/recurrent NPC.

1. EBV DNA is a molecular marker for NPC. We have reported that only 61% patients with local recurrence undergoing nasopharyngectomy had positive plasma EBV DNA. The sensitivity was lower in local recurrence compared with same stage in pretreatment NPC, 86% T1 versus 38% rT1. EBV DNA in nasopharyngeal brush has been reported to be 96% sensitive and 96% specific for NPC before treatment. EBV DNA in nasopharyngeal swab was reported to disappear after radiotherapy and re-appear with mucosal local recurrence with 100 % sensitivity and 98% specificity in a small case study of 11 patients with local recurrences, the results demonstrate its potential detection of local recurrences that are missed by our conventional follow-up. It however needs further prospective longitudinal study for verification.
2. Methylation of the CG rich promoter region of many tumor suppressor genes have been found to be a common genetic abnormality in NPC, but not in normal nasopharynx. We have shown that methylated promoter DNA are detectable in peripheral blood and nasopharyngeal swab of NPC patients, but rarely in normal controls. By using combination of 3 methylated genes in plasma, we have found 38% sensitive for detection of local recurrence.

2. Study objective To evaluate the sensitivity and specificity of the combination of EBV and methylation marker genes in body fluids of both plasma and nasopharyngeal brush together for screening of early salvageable local residual and recurrent NPC that are missed by conventional clinical follow-up protocol.

3. Hypothesis tested:

1. Patients in remission without residual or recurrent tumor after treatment should have persistently negative or very low background level of markers in both nasopharyngeal brush and plasma on follow-up.
2. Patients with residual or recurrent local or nodal tumors have either persistently high level of markers beyond 8th week or initial disappearance/reduction to very low background level followed by reappearance/increasing level of markers again on follow-up. The temporal change in quantity of markers is important to reflect the tumor load of residual and recurrent NPC before clinical presentation. We hypothesize that these pattern will be observed in those patients with residual/recurrent NPC at their early salvageable stages before clinical presentation.

4. Methodology of study:

1. Before treatment

   1. Nasopharyngeal brush of tumor is collected under endoscopic guidance.
   2. NPC biopsy specimen is then collected for histologic section and also freshly frozen in liquid nitrogen and stored in -80C freezer for subsequent study.
   3. 20ml EDTA blood is also collected for study.
   4. The EBV DNA and methylation markers will be screened in the tumor, nasopharyngeal brush and blood by using methylation specific quantitative PCR method. The laboratory protocols have been reported from our previous publications on EBV DNA and methylation studies.
2. Post-treatment reassessment of residual NPC

   1. Based on our published results on the study of time of remission of residual NPC after treatment, we have our routine follow-up protocol to perform endoscopic assessment and random biopsy of the nasopharynx at post-treatment 8th week for evaluation of residual NPC.
   2. At the time of endoscopy at 8th week, nasopharyngeal brush and 20 ml of blood will be collected for study of biomarkers. The EBV and specific methylation markers of the patient selected from patient's tumor biopsy findings will be used for each individual patient to screen residual NPC.
   3. Of those patients who have positive biopsy at 8th week, repeat biopsy will be done at 10th week. If the biopsy is still positive at 10th week, salvage treatment of either re-irradiation or nasopharyngectomy as appropriate will be arranged. If the repeat biopsy at 10th week becomes negative, the patient will be reassessed in 4 weeks.
   4. Of those patients with negative findings of both biomarkers and biopsy at 8th week, the patient will be followed-up according to schedule monthly.
   5. Of those patients who have positive biomarkers but negative biopsy at 8th week, further nasopharyngeal biopsies will be performed at 10th week to maker sure there is no missing of local residual NPC from the previous biopsy at 8th week. Radiologic imaging will also be performed at this time. The nasopharyngeal brush and blood tests will also be repeated to keep track of the temporal change with time. Patients who have positive biopsy at 10th week will be given appropriate salvage treatment of radiotherapy or surgery, and these patients are benefited by the molecular screening. Patients who have persistently negative biopsy at 10th week will be followed up according to schedule, and if they have no recurrence at follow-up, these patients have false positive molecular surveillance.
3. Subsequent follow-up for detection of recurrent NPC

   1. A patient who has negative post-treatment nasopharyngeal biopsy at 8th/10th week will be followed up every month in first year, every 2 months in second year and every 3 months in third - fifth year for total 5 years. It is expected that 11% of them in fact will subsequently develop local recurrence. It is our routine protocol to perform nasoendoscopy to examine the nasopharynx during each follow-up. If there is no suspicious lesion seen in the nasopharynx, biopsy will not be done and the patient will be rescheduled for follow-up.
   2. Nasopharyngeal biopsy will be taken if suspicious lesion is seen during follow-up endoscopy. If the biopsy is proven to be recurrence, the patient will be managed accordingly. If the biopsy is negative, the patient will be rescheduled for regular follow-up.
   3. Nasopharyngeal brush and 20 ml of blood will be collected at follow-up every 2 months for 1st and 2nd year and every 3 months in 3rd to 5th year for study.

      The EBV and specific methylation markers of the patient selected from patient's tumor biopsy findings will be reassessed for each individual patient to screen local recurrence.
   4. If a patient has negative nasoendoscopic finding and negative molecular biomarker findings in both plasma and nasopharyngeal brush, the patient will be regularly followed up as scheduled.
   5. If a patient has negative nasoendoscopic finding, but a positive molecular marker result is found in at least one of the body fluids or marker, the patient will be thoroughly reassessed for recurrence that are missed during routine clinical follow-up. The patient will have PET/CT/MRI imaging and random multiple nasopharyngeal biopsies to assess for possible local recurrence. Since a positive plasma finding may be due to nodal or distant metastasis, other sites of recurrence or new cancer will be investigated as judged necessary clinically. If the nasopharyngeal biopsy is positive or other site of recurrence is found, the patient will be managed by salvage treatment accordingly as appropriate. These patients are benefited by the molecular surveillance with true positive result. If the search for recurrence are all negative, the patient will be rescheduled for regular follow-up, and if the patient is proven no recurrence on further follow-up, the molecular surveillance is considered false positive.
4. End point of follow-up Post-treatment 5 years follow-up status will be our end point of study for each patient.
5. Number of patients recruited and recruitment criteria:

There are 130-150 new NPC patients annually in Queen Mary Hospital. We plan to recruit 350 patients for the longitudinal study starting from January 2006. The patients recruited should be medically fit for curative radiotherapy without distant metastasis before treatment. A total of 350 patients are expected to be recruited in 2008. Of these 350 patients, we expect to see about 35 patients who are found to have no residual local tumor with imaging and biopsy assessment at 8th week after radiotherapy with conventional follow-up, but subsequently develop isolated local recurrence within 5 years of follow-up. We would be able to know how many of these local recurrence will be benefited by early detection with molecular surveillance, their stage of recurrence and treatment outcome. Of these 350 patients, we expect to have about 20 patients with nodal recurrence.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with nasopharngeal carcinoma
* will receive radiotherapy after basline NP brush

Exclusion Criteria:

* has received radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nasopharngeeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of the combination of EBV and methylation marker genes in body fluids of both plasma and nasopharyngeal brush | 12 years

IPD SHARING:
Plan to Share IPD: Undecided